CLINICAL TRIAL: NCT04182711
Title: Feasibility Study of a Non-invasive Device to Quickly, Easily and Accurately Measure Respiration in a Clinical Setting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changi General Hospital (Other)
Collaborators: Agency for Science, Technology and Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1
Record Dates: First submitted 2019-11-27; First posted 2019-12-02 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: COPD
Keywords: COPD; Asthma; Pneumonia; Congestive heart failure
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma; Pneumonia; Heart Failure | interventions — Equipment and Supplies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Device Arm (Experimental): The aim in the 1st phase is to benchmark the device against manual counting of respiration (number of breaths per minute). The aim in the 2nd phase is to benchmark the device against existing technologies, namely lead-based-ECG sensing, acoustic sensing and capnography. This phase can have a mix of patients having either COPD, asthma, pneumonia or any other respiratory diseases
  Interventions: Device: Device

INTERVENTIONS:
Device: Device — Phase 1: Time taken for each patient is 25 mins Phase 2: Time taken for each patient is 30 mins

SUMMARY:
Healthcare facilities worldwide still measure respiration manually by counting and timing chest movements. In clinical departments that are fast-paced in nature and that have either high patient volumes or require more accurate measurements (e.g. emergency and respiratory wards), manual methods of counting respiration can be slow, laborious and highly subjective. While potential solutions such as electrocardiography (ECG) and capnography (CPG) have been explored for more objective monitoring of respiration, they are not fast enough due to long setup times to get patient and system ready and prolonged periods of connection to patients. Furthermore, such ECG/CPG based solutions can be costly, are generally sufficient for patients in high dependency units, and may be impractical to deploy in a remote setting.

DETAILED DESCRIPTION:
The study will be divided into 2 phases - 1st phase will last 1.5 months and will aim to recruit at least 50 patients and at most 100 patients. This phase will aim to recruit near-equal split of patients across the 3 disease states of COPD, asthma and pneumonia - 35 COPD, 35 Asthma and 30 pneumonia patients. The 2nd phase will last 3 months and will aim to recruit at least 50 patients. This phase can have a mix of patients having either COPD, asthma, pneumonia, congestive heart failure or any other respiratory diseases

The aim in the 1st phase is to benchmark the device against manual counting of respiration (number of breaths per minute). The aim in the 2nd phase is to benchmark the device against existing technologies, namely lead-based-ECG sensing, acoustic sensing and capnography. This phase can have a mix of patients having either COPD, asthma, pneumonia or any other respiratory diseases

Following is the study protocol that will be implemented over the 2 phases:

Phase 1: 1.5 months - 100 patients - General Wards (Time taken for each patient is 25 mins)

a. Delegated study team members will brief the study details to the potential participants. Investigators will answer the query from potential participants if any, and complete the consent process. (5 mins) b. Trial coordinator will setup the device as follows: (10 mins) i. Disinfect the device by wiping with an alcohol swab, ii. Turn on the sensor - ensure the USB dongle is connected to the RIGHT ports on the laptop - check that the USB dongle AND the sensor light is NOT blinking iii. Paste the sensor on patient using a medical-grade adhesive tape.

c. Trial coordinator will begin data collection by double click the software .exe file - select the COM ports and enter participant no. (a folder will be created in root directory for the participant number) d. Click "run" button on the software and start to manually count the number of breaths after 1 minute. After 1 minute, the number of breaths counted manually will be recorded on the case report form.4 rounds of 1-minute measurements will be taken e. Trial coordinator will turn off the device and pass it back to team-member or keep it. Trial coordinator will remove the medical-grade adhesive tape and throw it away. (5 mins) f. Team-member will post-process the collected respiration data, benchmark against the manually counted data in the data collection form provided by trial coordinator and discuss the results with investigating P.Is.

Phase 2: 3 months - 50 patients - Medical intensive care units (MICU), medical dependency units (MDU), cardiology high dependency units, and general wards (for congestive heart failure patients) (Time taken for each patient is 30 mins) g. Delegated study team members will brief the study details to the potential participants. Investigators will answer the query from potential participants if any, and complete the consent process. In the event that the patient is unable to provide consent, the next-of-kin will be approached for consent. (5 mins) h. Trial coordinator will setup the device as follows: (10 mins) i. Disinfect the device by wiping with an alcohol swab, ii. Turn on the sensor - ensure the USB dongle is connected to the RIGHT ports on the laptop - check that the USB dongle AND the sensor light is NOT blinking iii. Paste the sensor on patient using a medical-grade adhesive tape. iv. Attach another sensor on the patient's finger using an adapter. The purpose of this is to collect heart rate and Sp02, and to calculate respiration from the collected data.

i. Trial coordinator will begin data collection by double click the software .exe file - select the COM ports and enter participant no. (a folder will be created in root directory for the participant number) j. Click "run" button on the software. After 1 minute, the number of breaths, heart rate and Sp02 from other technology devices will be recorded on the case report form.4 rounds of 1-minute measurements will be taken.

k. Trial coordinator will turn off the device and pass it back to team-member or keep it. Trial coordinator will remove the medical-grade adhesive tape and throw it away. (5 mins). Trial coordinator will also remove the device and adapter from the finger location.

l. Team-member will post-process the collected respiration data, benchmark it and discuss the results with investigating P.Is.

All data collected will be anonymous and no video-taping will be done. The trial coordinator will act as the control arm. They will measure the respiration or breathing rate of the subject manually - by counting the number of breaths per minute. The non-control arm will be the device itself and it will be benchmarked to the manual respiration data collected by the trial coordinator. The data collected will be kept with the P.I and confidentially of the data will strictly be maintained. The case report forms or the collection forms will be passed to the P.I. and kept safely. The subject may choose to withdraw from the study at any time.

The device is based on multi-modal sensing using illumination at extremely low emission levels on the order of microwatts. This sensing technique is able to detect the micro-vibrations along the neck due to breathing.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with cardio-respiratory diseases of either asthma, COPD, pneumonia, congestive heart failure or any other respiratory diseases.
* Patients should be able to provide informed consent either personally or through the next-of-kin. The study will consider a mix of mild to severe cases and will not be specific to either gender, sex or ethnicity.
* Patients with congestive heart failure only from general ward or cardiology high dependency units.

Exclusion Criteria:

* Patients that are either mentally incompetent, younger than 21 years of age, prisoners, pregnant or breastfeeding women.
* Patients with metallic/electrical implants e.g. pacemakers, cardiac devices, airway stents, neurostimulators etc.
* Patients with coronary stents insitu are eligible for enrolment into the study. Any medical condition which makes the candidate an inappropriate subject for study participation, in the investigator's judgment will further be excluded.
* Congestive heart failure patients on antibiotics or with infection.
* Congestive heart failure patients beyond 72 hours of presentation from enrolment. Intent is to capture congestive heart failure at the acute stage, prior to resolving.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Accuracy of this device on disease subjects in a clinical setting. | 4.5 Months
  The device will be compared against "gold-standard" manual counting and against existing technologies such as lead-based ECG, capnography and acoustic-based sensing.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Augustine Tee, Principal Investigator — Changi General Hospital
Locations (1):
- Clinical Trials & Research Unit, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No